CLINICAL TRIAL: NCT01833702
Title: Use of a Mobile-based Pain Assessment Application for SCD Patients
Brief Title: Use of a Mobile-based App for SCD Patients
Acronym: SMART
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00037857
Record Dates: First submitted 2013-04-13; First posted 2013-04-17 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2018-11

CONDITIONS: Sickle Cell Disease; Chronic Pain
Keywords: Sickle cell; Pain
MeSH Terms: conditions — Anemia, Sickle Cell; Chronic Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Automated response: Canned responses are provided at the end of daily entries
- No automated feedback: Canned responses are not provided at the end of daily entries

SUMMARY:
The study will seek to enroll 100 sickle cell or thalassemia patients who are age 12 or older who have access to a smartphone or tablet with Internet access daily.

The study will evaluate patient-reported comfort level with using a mobile device to record their pain levels, as well as adherence to recording these levels daily.

The study will track patients' assessment of their pain, actions taken, and outcomes related to pain management and provider involvement.

This study will attempt to collect information about differences in the use of two traditional pain assessment modes (verbal scale and paper) versus the use of a pain assessment tool on a mobile device in the form of a smartphone, tablet, or iPad with an Android or iOS operating system.

DETAILED DESCRIPTION:
The study will evaluate patient-reported comfort level with using a mobile device to record their pain levels, as well as adherence to recording these levels daily. The study will track patients' assessment of their pain, actions taken, and outcomes related to pain management and provider involvement. This study will attempt to collect information about differences in the use of two traditional pain assessment modes (verbal scale and paper) versus the use of a pain assessment tool on a mobile device in the form of a smartphone, tablet, or iPad with an Android or iOS operating system. The study will seek to enroll 100 sickle cell or thalassemia patients who are age 12 or older who have access to a smartphone or tablet with Internet access daily. Patients enrolled in this study will be ask to use a mobile device such as a smartphone or a tablet with Android or iOS operating system to record daily pain level and related information once daily or more frequently for a period of forty-two days. A 1:1 randomization assignment will be made to have patients receive automated "canned" provider feedback or not.

ELIGIBILITY:
Inclusion Criteria:

* SCD, thalassemia, or history of experiencing pain

Exclusion Criteria:

* none

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients experiencing pain or patients with sickle cell disease
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Usability | 42 days
  Patients are able to use a mobile device to record daily symptoms, including pain, and interventions, including medication administration.

CONTACTS AND LOCATIONS:
Overall Officials: Jude Jonassaint, RN, Principal Investigator — Duke University; Laura De Castro, MD, Principal Investigator — Duke University; Nirmish Shah, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States